CLINICAL TRIAL: NCT05992688
Title: The Sweet Kids Study (Stevia on Weight and Energy Effect Over Time)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: Cargill (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 275844
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Adiposity; Insulin Sensitivity; Weight Gain; Blood Pressure; Lipoproteins
Keywords: Cardiometabolic health
MeSH Terms: conditions — Obesity; Insulin Resistance; Weight Gain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sucrose sweetened beverage (Active Comparator): Sucrose (i.e. sugar): 31.2 g sugar (124.8 Kcal per serving). Participants will be asked to consume the study product once a day for 8 to 14 weeks if they have normal weight or excessive weight, respectively.
  Interventions: Other: Sucrose sweetened beverage
- Stevia sweetened beverage (Experimental): The stevia-sweetened beverage contains 48.6 mg of steviol equivalents. Participants will be asked to consume the study product once a day for 8 to 14 weeks if they have normal weight or excessive weight, respectively.
  Interventions: Other: Stevia sweetened beverages
- Calorie free flavored water beverage (Active Comparator): Flavored water. Participants will be asked to consume the study product once a day for 8 to 14 weeks if they have normal weight or excessive weight, respectively.
  Interventions: Other: Calorie free flavored water beverage

INTERVENTIONS:
Other: Sucrose sweetened beverage — Children who habitually consume sugar (sucrose) - sweetened beverages who are randomized to this arm, will consume the study product for 8 to 14 weeks.
  Arms: Sucrose sweetened beverage
Other: Stevia sweetened beverages — Children who habitually consume sugar (sucrose) - sweetened beverages who are randomized to this arm, will consume the study product for 8 to 14 weeks.
  Arms: Stevia sweetened beverage
Other: Calorie free flavored water beverage — Children who habitually consume sugar (sucrose) - sweetened beverages who are randomized to this arm, will consume the study product for 8 to 14 weeks.
  Arms: Calorie free flavored water beverage

SUMMARY:
This is an 8 to14-week three-arm randomized controlled in children 8 to 12 years old.

The main purpose of the study is to evaluate if stevia has benefits for weight control and metabolic function relative to caloric sweeteners, and whether it provides benefits in this regard similar to water.

DETAILED DESCRIPTION:
Up to 150 children will be enrolled in the study to achieve a final sample of 90 completers (30 per group). The proposed study will be an 8 to 14-week, three-arm, randomized, controlled, blinded trial in children ages 8 to 12 years from the Central Arkansas region. Children will be randomized to consume one of three beverages: 1) sucrose-sweetened beverage, 2) stevia-sweetened beverage, or 3) calorie-free flavored water beverage. Participants with excessive weight (BMI percentile ≥85th and <140 percent of the 95th percentile) will complete a 14-week intervention whereas normal-weight (BMI percentile <85th) participants will complete an 8-week intervention in parallel.

ELIGIBILITY:
Inclusion Criteria

* Age 8-12 years
* Normal weight: BMI percentile ≥5th to <85th
* Excessive weight: BMI percentile ≥ 85th and <140% of the 95th percentile or BMI ≥35 to <40 kg/m2
* Current consumption of sugar sweetened beverages (≥2 times /wk)
* Low consumption of non-nutritive sweeteners (≤ 3 time/wk)
* Willingness to consume experimental products Exclusion Criteria
* Children with class 3 obesity (i.e., BMI ≥ 140% of the 95th percentile or BMI ≥ 40.0 kg/m2)
* Dislike of experimental beverage taste (assessed at initial visit)
* Asthma that requires daily use of inhalers to keep symptoms under control.
* Asthma that requires use of rescue inhalers (e.g., albuterol) >2 days per week
* Exercise induced asthma.
* Autism spectrum disorder (e.g., Autistic disorder, Rett disorder, Asperger disorder, childhood disintegrative disorder, pervasive developmental disorder not otherwise specified (PDD-NOS).
* Attention deficit hyperactivity disorder (ADHD) currently under medication.
* Oppositional defiant disorder (ODD).
* Epilepsy.
* Cancer.
* Chronic kidney disease.
* Endocrine disorder (e.g., hypothyroidism and growth hormone deficiency).
* Autoimmune diseases (e.g., lupus, thyroiditis, juvenile idiopathic arthritis)
* Bleeding disorders (e.g., hemophilia)
* Chronic infections (e.g., HIV, hepatitis B, hepatitis C).
* Mental health disorders (e.g., depression and anxiety).
* Type 2 and type 1 diabetes mellitus.
* Other pre-existing medical conditions or medications as determined by the investigators to affect the outcomes of interest.
* If, during the screening or consent process, the parent or child expresses refusal to have blood drawn. However, participants may remain in the study if after initially agreeing to the blood draw and enrolling they change their minds and choose not to allow blood draws or if blood draws are unsuccessful.
* Dislike of study products assessed at initial visit.
* Fasting glucose ≥126 mg/dl at enrollment.
* Fasting A1C ≥6.5% at enrollment
* Less than 2 months since completion of antibiotics

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Body mass index (BMI) z-scores | Measurements will be obtained at enrollment (baseline) and again at weeks 4 and 8 for all participants. Children with excessive weight will also complete an additional assessment at week 14.
  The change in BMI z-score will be calculated: BMI z-score at completion of the study minus BMI z-score at baseline
Fat mass index z-scores | Measurements will be obtained at enrollment (baseline) and again at weeks 4 and 8 for all participants. Children with excessive weight will also complete an additional assessment at week 14.
  The change in fat mass index (FMI) z-score will be calculated: FMI z-score at completion of the study minus FMI z-score at baseline.
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | Measurements will be obtained at enrollment (baseline) and again at weeks 4 and 8 for all participants. Children with excessive weight will also complete an additional assessment at week 14.
  HOMA-IR is a unitless estimate of insulin resistance, and it is calculated from fasting glucose and insulin
Fasting plasma lipids (Total cholesterol, HDL-cholesterol, triglycerides, LDL-cholesterol) | Measurements will be obtained at enrollment (baseline) and again at weeks 4 and 8 for all participants. Children with excessive weight will also complete an additional assessment at week 14.
  Fasting plasma lipids, mg/dl
Blood pressure percentiles | Measurements will be obtained at enrollment (baseline) and again at weeks 4 and 8 for all participants. Children with excessive weight will also complete an additional assessment at week 14.
  Systolic and diastolic blood pressure percentiles calculated using reference standards from the American Academy of Pediatrics.

SECONDARY OUTCOMES:
Gut microbial communities | Measurements will be obtained at enrollment (baseline) and again at week 8 for all participants. Children with excessive weight will also complete an additional assessment at week 14.
  Shift in gut microbial communities will be assessed using 16S analyses

CONTACTS AND LOCATIONS:
Overall Officials: Eva Diaz, M.D., Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
All study subject materials will be assigned a unique identifying code or number. The key to the code will be kept in a shared network folder with access granted only to study staff who have had appropriate CITI training. Only study investigators/staff will have access to the code and information that identifies the subject in this study. Coded data for all primary and secondary outcomes as well as secondary data analysis will be shared with the Sponsor (Cargill Corporation) using an approved shared folder .